CLINICAL TRIAL: NCT05382104
Title: A Phase 1, Open-Label, Randomized, Crossover Study to Evaluate the Effect of Food on Maribavir (TAK-620) Pharmacokinetics in Healthy Adult Participants
Brief Title: Maribavir Food-Effect Study in Healthy Adults Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TAK-620-1025
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Results first posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — maribavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Sequence 1: Treatment A + Treatment B + Treatment C (Experimental): Participants will receive maribavir single 400 mg tablet, on Day 1 of Period 1 under fasting condition (Treatment A), followed by maribavir single 400 mg tablet, on Day 1 of Period 2. administered with a low fat/low calorie meal (Treatment B), and further followed by maribavir single 400 mg tablet, on Day 1 of Period 3 administered with a high fat/high calorie meal (Treatment C). There will be a washout period of minimum of 72 hours between each ID dosing.
  Interventions: Drug: Maribavir
- Sequence 2: Treatment A + Treatment C + Treatment B (Experimental): Participants will receive maribavir single 400 mg tablet, on Day 1 of Period 1 under fasting condition (Treatment A), followed by maribavir single 400 mg tablet on Day 1 of Period 2 administered with a high fat/high calorie meal (Treatment C), and followed by maribavir single 400 mg tablet, on Day 1 of Period 3 administered with a low fat/low calorie meal (Treatment B). There will be a washout period of minimum of 72 hours between each ID dosing.
  Interventions: Drug: Maribavir
- Sequence 3: Treatment B + Treatment A + Treatment C (Experimental): Participants will receive maribavir single 400 mg tablet, on Day 1 of Period 1 administered with a low fat/low calorie meal (Treatment B), followed by maribavir single 400 mg tablet, on Day 1 of Period 2 under fasting condition (Treatment A), and followed by maribavir single 400 mg tablet, on Day 1 of Period 3 administered with a high fat/high calorie meal (Treatment C). There will be a washout period of minimum of 72 hours between each ID dosing.
  Interventions: Drug: Maribavir
- Sequence 4: Treatment B + Treatment C + Treatment A (Experimental): Participants will receive maribavir single 400 mg tablet, on Day 1 of Period 1 administered with a low fat/low calorie meal (Treatment B), followed by maribavir single 400 mg tablet, on Day 1 of Period 2 administered with a high fat/high calorie meal (Treatment C), and followed by maribavir single 400 mg tablet, on Day 1 of Period 3 under fasting condition (Treatment A). There will be a washout period of minimum of 72 hours between each ID dosing.
  Interventions: Drug: Maribavir
- Sequence 5: Treatment C + Treatment A + Treatment B (Experimental): Participants will receive maribavir single 400 mg tablet, on Day 1 of Period 1 administered with a high fat/high calorie meal (Treatment C), followed by maribavir single 400 mg tablet, on Day 1 of Period 2 under fasting condition (Treatment A), and followed by maribavir single 400 mg tablet, on Day 1 of Period 3 administered with a low fat/low calorie meal (Treatment B). There will be a washout period of minimum of 72 hours between each ID dosing.
  Interventions: Drug: Maribavir
- Sequence 6: Treatment C + Treatment B + Treatment A (Experimental): Participants will receive maribavir single 400 mg tablet, on Day 1 of Period 1 administered with a high fat/high calorie meal (Treatment C), followed by maribavir single 400 mg tablet, on Day 1 of Period 2 administered with a low fat/low calorie meal (Treatment B), and followed by maribavir single 400 mg tablet on Day 1 of Period 3 under fasting condition (Treatment A). There will be a washout period of minimum of 72 hours between each ID dosing.
  Interventions: Drug: Maribavir

INTERVENTIONS:
Drug: Maribavir — Maribavir single 400 mg tablet under three different food conditions (fasted, low fat/low calorie meal, and high fat/high calorie meal) depending upon the treatment sequence allocation on Day 1 of each treatment period.
  Other Names: TAK-620

SUMMARY:
The main goals of this study are: 1) To assess the relative bioavailability of a single oral dose of 400 mg maribavir commercial (marketed) tablet formulation administered with a low-fat/low-calorie meal relative to administration under fasting conditions. 2) To assess the relative bioavailability of a single oral dose of 400 mg maribavir commercial (marketed) tablet formulation administered with a high-fat/high calorie meal relative to administration under fasting conditions.

A single dose of 400 mg maribavir (commercial [marketed] tablet formulation) will be administered orally under 3 different feeding conditions:

1. Fasting (Treatment A),
2. Fed following a low-fat/low-calorie meal (Treatment B), and
3. Fed following a high fat/high-calorie meal (Treatment C).

There will be a washout period of a minimum of 72 hours between each single dose of investigational drug (ID) administration on Day 1 in each treatment cycle of 3 days.

Pharmacokinetic samples will be collected at pre-dose and up to 36 hours post-dose in each treatment period.

Safety and tolerability will be assessed throughout the study by Treatment Emergent Adverse Events (TEAEs), vital signs, electrocardiograms (ECGs), and clinical laboratory evaluations.

ELIGIBILITY:
Inclusion Criteria

Participants must fulfill the following inclusion criteria before the first dose of the Investigational drug (ID) to be eligible for participation in the study:

* An understanding, ability, and willingness to fully comply with study procedures and restrictions and ability to voluntarily provide written, signed, and dated (personally or via a legally authorized representative) informed consent
* Age 19-55 years, inclusive at the time of consent, at the screening visit.
* Male, or non-pregnant, non-breastfeeding female who agrees to comply with any applicable contraceptive requirements of the protocol or female of non-childbearing potential.
* Healthy as determined by the Investigator or designee on the basis of screening evaluations and medical history.
* Hemoglobin for males greater than or equal to (>=) 135.0 gram per liter (g/L) and females >=120.0 g/L at the screening visit and on Day 1 of Treatment Period 1.
* Body mass index (BMI) between 18.0 and 30.0 kilogram per square meter (kg/m^2), inclusive with a body weight greater than (>) 50 kilogram (kg) (110 pound [lbs]), at the screening visit.
* Ability to swallow a dose of the ID.

Exclusion Criteria

Participants must not be enrolled in the study if they meet any of the following criteria before the first dose of the ID:

* History or presence of gastritis, Gastrointestinal (GI) tract, hepatic disorder or cholecystectomy, history of treated or untreated Helicobacter pylori, ulcer disease or other clinical GI condition and history of any hematological, hepatic, respiratory, cardiovascular, renal, neurological or psychiatric disease, gall bladder removal, or current recurrent disease that could affect the action, absorption, or disposition of the ID, or clinical or laboratory assessments.
* Current or relevant history of physical or psychiatric illness, any medical disorder that may require treatment or make the participant unlikely to fully complete the study, or any condition that presents undue risk from the ID or procedures.
* Known or suspected intolerance or hypersensitivity to the ID, closely related compounds, or any of the stated ingredients and excipients.
* Significant illness, as judged by the Investigator or designee, within 2 weeks of the first dose of the ID.
* Has diarrhea within 4 hours of the first dose of the ID.
* Donors of blood or blood products (e.g., plasma or platelets) within 60 days prior to receiving the first dose of the ID.
* Within 30 days prior to the first dose of the ID:

  * Have used any investigational product (if elimination half-life is less than [<] 6 days, otherwise 5 half-lives).
  * Have been enrolled in a clinical study (including vaccine studies) that may impact this study.
  * Have had any substantial changes in eating habits.
* Systolic blood pressure >140 millimeters of mercury (mmHg) or <90 mmHg, and diastolic blood pressure >90 mmHg or <50 mmHg, at the screening visit.
* Twelve-lead ECG with corrected QT interval (QTc) >450 millisecond (msec) at the screening visit.
* Known history of alcohol or other substance abuse within the last year.
* Male participants who consume more than 21 units of alcohol per week or 3 units per day. Female participants who consume more than 14 units of alcohol per week or 2 units per day.
* A positive screen for alcohol or drugs of abuse at the screening visit or on Day -1 of Treatment Period 1.
* A positive human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), or Hepatitis C virus (HCV) antibody screen at the screening visit.
* Use of tobacco in any form or other nicotine-containing products in any form. Ex-users must self-report that they have stopped using tobacco for at least 3 months prior to receiving the first dose of the ID.
* Routine consumption of more than 2 units of caffeine per day or participants who experience caffeine withdrawal headaches. Decaffeinated coffee, tea, or cola are not considered to contain caffeine.
* Current use of any prescription medication with the exception of hormonal contraceptives and hormonal replacement therapy.
* Current use of antacids, proton pump inhibitors, or H2 antagonists within 14 days of the first dose of the ID.
* Inability or unwillingness to consume 100 percent of high-fat meal or low-fat meal (including participants with lactose or gluten intolerance).
* Recent history (within 1 month) of oral/nasal cavity infections, history of gastroesophageal reflux, asthma treatment with albuterol, or zinc supplementation.
* Participants with dry mouth syndrome or burning mouth syndrome or participants suffering from dysgeusia.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-07-02 (Actual); Study Completion 2022-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/256f7e94e98d41f6?idFilter=%5B%22TAK-620-1025%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at single center in the United States from 25 May 2022 to 02 July 2022.
Pre-assignment Details: A total of 31 healthy participants were enrolled in this 3-period crossover study and were randomized to 1 of 6 treatment sequences to receive maribavir 400 milligrams (mg) tablet in fasting state (Treatment A), fed following a low-fat/low-calorie meal (Treatment B) or fed following a high-fat/high-calorie meal (Treatment C).
Groups:
- Sequence 1: Treatment A + Treatment B + Treatment C: Participants received maribavir single 400 mg tablet, on Day 1 of Treatment Period 1 under fasting condition (Treatment A), followed by maribavir single 400 mg tablet, on Day 1 of Treatment Period 2 administered with a low fat/low calorie meal (Treatment B), and further followed by maribavir single 400 mg tablet, on Day 1 of Treatment Period 3 administered with a high fat/high calorie meal (Treatment C). A washout period of minimum of 72 hours between each investigational drug (ID) dosing was maintained.
- Sequence 2: Treatment A + Treatment C + Treatment B: Participants received maribavir single 400 mg tablet, on Day 1 of Treatment Period 1 under fasting condition (Treatment A), followed by maribavir single 400 mg tablet, on Day 1 of Treatment Period 2 administered with a high fat/high calorie meal (Treatment C), and followed by maribavir single 400 mg tablet, on Day 1 of Treatment Period 3 administered with a low fat/low calorie meal (Treatment B). A washout period of minimum of 72 hours between each ID dosing was maintained.
- Sequence 3: Treatment B + Treatment A + Treatment C: Participants received maribavir single 400 mg tablet, on Day 1 of Treatment Period 1 administered with a low fat/low calorie meal (Treatment B), followed by maribavir single 400 mg tablet, on Day 1 of Treatment Period 2 under fasting condition (Treatment A), and followed by maribavir single 400 mg tablet, on Day 1 of Treatment Period 3 administered with a high fat/high calorie meal (Treatment C). A washout period of minimum of 72 hours between each ID dosing was maintained.
- Sequence 4: Treatment B + Treatment C + Treatment A: Participants received maribavir single 400 mg tablet, on Day 1 of Treatment Period 1 administered with a low fat/low calorie meal (Treatment B), followed by maribavir single 400 mg tablet, on Day 1 of Treatment Period 2 administered with a high fat/high calorie meal (Treatment C), and followed by maribavir single 400 mg tablet, on Day 1 of Treatment Period 3 under fasting condition (Treatment A). A washout period of minimum of 72 hours between each ID dosing was maintained.
- Sequence 5: Treatment C + Treatment A + Treatment B: Participants received maribavir single 400 mg tablet, on Day 1 of Treatment Period 1 administered with a high fat/high calorie meal (Treatment C), followed by maribavir single 400 mg tablet, on Day 1 of Treatment Period 2 under fasting condition (Treatment A), and followed by maribavir single 400 mg tablet, on Day 1 of Treatment Period 3 administered with a low fat/low calorie meal (Treatment B). A washout period of minimum of 72 hours between each ID dosing was maintained.
- Sequence 6: Treatment C + Treatment B + Treatment A: Participants received maribavir single 400 mg tablet, on Day 1 of Treatment Period 1 administered with a high fat/high calorie meal (Treatment C), followed by maribavir single 400 mg tablet, on Day 1 of Treatment Period 2 administered with a low fat/low calorie meal (Treatment B), and followed by maribavir single 400 mg tablet, on Day 1 of Treatment Period 3 under fasting condition (Treatment A). A washout period of minimum of 72 hours between each ID dosing was maintained.
Period: Period 1 (2 Days)
Arm/Group | Sequence 1: Treatment A + Treatment B + Treatment C | Sequence 2: Treatment A + Treatment C + Treatment B | Sequence 3: Treatment B + Treatment A + Treatment C | Sequence 4: Treatment B + Treatment C + Treatment A | Sequence 5: Treatment C + Treatment A + Treatment B | Sequence 6: Treatment C + Treatment B + Treatment A
Started | 5 | 6 | 5 | 5 | 5 | 5
Completed | 5 | 6 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1 (72 Hours)
Arm/Group | Sequence 1: Treatment A + Treatment B + Treatment C | Sequence 2: Treatment A + Treatment C + Treatment B | Sequence 3: Treatment B + Treatment A + Treatment C | Sequence 4: Treatment B + Treatment C + Treatment A | Sequence 5: Treatment C + Treatment A + Treatment B | Sequence 6: Treatment C + Treatment B + Treatment A
Started | 5 | 6 | 5 | 5 | 5 | 5
Completed | 5 | 6 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 (2 Days)
Arm/Group | Sequence 1: Treatment A + Treatment B + Treatment C | Sequence 2: Treatment A + Treatment C + Treatment B | Sequence 3: Treatment B + Treatment A + Treatment C | Sequence 4: Treatment B + Treatment C + Treatment A | Sequence 5: Treatment C + Treatment A + Treatment B | Sequence 6: Treatment C + Treatment B + Treatment A
Started | 5 | 6 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Period: Washout Period 2 (72 Hours)
Arm/Group | Sequence 1: Treatment A + Treatment B + Treatment C | Sequence 2: Treatment A + Treatment C + Treatment B | Sequence 3: Treatment B + Treatment A + Treatment C | Sequence 4: Treatment B + Treatment C + Treatment A | Sequence 5: Treatment C + Treatment A + Treatment B | Sequence 6: Treatment C + Treatment B + Treatment A
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3 (2 Days)
Arm/Group | Sequence 1: Treatment A + Treatment B + Treatment C | Sequence 2: Treatment A + Treatment C + Treatment B | Sequence 3: Treatment B + Treatment A + Treatment C | Sequence 4: Treatment B + Treatment C + Treatment A | Sequence 5: Treatment C + Treatment A + Treatment B | Sequence 6: Treatment C + Treatment B + Treatment A
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety set included all participants who received at least 1 dose of maribavir.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1: Treatment A + Treatment B + Treatment C | Sequence 2: Treatment A + Treatment C + Treatment B | Sequence 3: Treatment B + Treatment A + Treatment C | Sequence 4: Treatment B + Treatment C + Treatment A | Sequence 5: Treatment C + Treatment A + Treatment B | Sequence 6: Treatment C + Treatment B + Treatment A | Total
Number analyzed (Participants) | 5 | 6 | 5 | 5 | 5 | 5 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (5.02) | 37.7 (6.35) | 26.0 (5.61) | 37.2 (11.48) | 39.2 (7.92) | 42.8 (10.26) | 35.2 (9.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 2 | 1 | 2 | 10
  Male | 3 | 5 | 3 | 3 | 4 | 3 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 5 | 4 | 5 | 5 | 5 | 5 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 5 | 1 | 3 | 1 | 17
  White | 1 | 3 | 0 | 4 | 2 | 4 | 14
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Maribavir
Description: Cmax of maribavir in plasma was reported using the non-compartmental analysis.
Time Frame: Day 1: Pre dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24 and 36-hours post-dose
Population: The pharmacokinetic (PK) set included all participants who received at least 1 dose of maribavir, did not vomit or had diarrhea within 4 hours of the ID dosing, and had 5 or more post-dose time points with evaluable post-dose maribavir concentration values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Groups:
- Treatment A: Maribavir 400 mg: Participants received maribavir single 400 mg tablet, under fasted conditions on Day 1 of Treatment Period 1, 2 and 3.
- Treatment B: Maribavir 400 mg: Participants received maribavir single 400 mg tablet, after low-fat/low-calorie meal on Day 1 of Treatment Period 1, 2 and 3.
- Treatment C: Maribavir 400 mg: Participants received maribavir single 400 mg tablet, after high-fat/high-calorie meal on Day 1 of Treatment Period 1, 2 and 3.
Arm/Group | Treatment A: Maribavir 400 mg | Treatment B: Maribavir 400 mg | Treatment C: Maribavir 400 mg
Number analyzed (Participants) | 30 | 29 | 30
microgram per milliliter (mcg/mL) | 17.8 (28.9) | 13.4 (23.3) | 12.7 (21.0)
Statistical Analysis 1: Comparison: Treatment A: Maribavir 400 mg vs Treatment B: Maribavir 400 mg; Test type: Equivalence — A linear mixed-effects model was applied to natural log (ln)-transformed Cmax with treatment, period, and sequence as fixed effects, and participant within sequence as a random effect. Point estimates and their associated 90 percent (%) confidence intervals (CIs) was constructed for the differences between Treatment B versus Treatment A. The point estimates and their associated 90% CIs were then back transformed to provide point estimates and 90% CIs for ratios of Treatment B versus Treatment A; Geometric Mean Ratio (%) = 76.62, 90% CI 2-sided [71.78 to 81.78] — Geometric mean ratio (%) was calculated as 100*(Treatment B / Treatment A)
Statistical Analysis 2: Comparison: Treatment A: Maribavir 400 mg vs Treatment C: Maribavir 400 mg; Test type: Equivalence — A linear mixed-effects model was applied to ln-transformed Cmax with treatment, period, and sequence as fixed effects, and participant within sequence as a random effect. Point estimates and their associated 90% CIs was constructed for differences between Treatment C versus Treatment A. The point estimates and their associated 90% CIs were then back transformed to provide point estimates and 90% CIs for ratios of Treatment C versus Treatment A; Geometric Mean Ratio (%) = 71.61, 90% CI 2-sided [67.14 to 76.37] — Geometric mean ratio (%) was calculated as 100*(Treatment C / Treatment A)

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve From the Time of Dosing to the Last Measurable Concentration (AUClast) of Maribavir
Description: AUClast of maribavir in plasma was reported using the non-compartmental analysis.
Time Frame: Day 1: Pre dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24 and 36-hours post-dose
Population: The PK set included all participants who received at least 1 dose of maribavir, did not vomit or had diarrhea within 4 hours of the ID dosing, and had 5 or more post-dose time points with evaluable post-dose maribavir concentration values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter(mcg*hr/mL)
Arm/Group | Treatment A: Maribavir 400 mg | Treatment B: Maribavir 400 mg | Treatment C: Maribavir 400 mg
Number analyzed (Participants) | 30 | 29 | 30
microgram*hour per milliliter(mcg*hr/mL) | 103 (30.0) | 85.6 (34.0) | 90.0 (33.2)
Statistical Analysis 1: Comparison: Treatment A: Maribavir 400 mg vs Treatment B: Maribavir 400 mg; Test type: Equivalence — A linear mixed-effects model was applied to ln-transformed AUClast with treatment, period, and sequence as fixed effects, and participant within sequence as a random effect. Point estimates and their associated 90% CIs was constructed for the differences between Treatment B versus Treatment A. The point estimates and their associated 90% CIs were then back transformed to provide point estimates and 90% CIs for ratios of Treatment B versus Treatment A; Geometric Mean Ratio (%) = 84.13, 90% CI 2-sided [80.74 to 87.66] — Geometric mean ratio (%) was calculated as 100*(Treatment B / Treatment A)
Statistical Analysis 2: Comparison: Treatment A: Maribavir 400 mg vs Treatment C: Maribavir 400 mg; Test type: Equivalence — A linear mixed-effects model was applied to ln-transformed AUClast with treatment, period, and sequence as fixed effects, and participant within sequence as a random effect. Point estimates and their associated 90% CIs was constructed for differences between Treatment C versus Treatment A. The point estimates and their associated 90% CIs were then back transformed to provide point estimates and 90% CIs for ratios of Treatment C versus Treatment A; Geometric Mean Ratio (%) = 87.35, 90% CI 2-sided [83.87 to 90.96] — Geometric mean ratio (%) was calculated as 100*(Treatment C / Treatment A)

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC0-infinity) of Maribavir
Description: AUC0-infinity of maribavir in plasma was reported using the non-compartmental analysis.
Time Frame: Day 1: Pre dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24 and 36-hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*hr/mL
Arm/Group | Treatment A: Maribavir 400 mg | Treatment B: Maribavir 400 mg | Treatment C: Maribavir 400 mg
Number analyzed (Participants) | 30 | 29 | 30
mcg*hr/mL | 106 (29.6) | 88.7 (34.3) | 93.2 (33.4)
Statistical Analysis 1: Comparison: Treatment A: Maribavir 400 mg vs Treatment B: Maribavir 400 mg; Test type: Equivalence — A linear mixed-effects model was applied to ln-transformed AUC0-infinity with treatment, period, and sequence as fixed effects, and participant within sequence as a random effect. Point estimates and their associated 90% CIs was constructed for the differences between Treatment B versus Treatment A. The point estimates and their associated 90% CIs were then back transformed to provide point estimates and 90% CIs for ratios of Treatment B versus Treatment A; Geometric Mean Ratio (%) = 84.74, 90% CI 2-sided [81.28 to 88.34] — Geometric mean ratio (%) was calculated as 100*(Treatment B / Treatment A)
Statistical Analysis 2: Comparison: Treatment A: Maribavir 400 mg vs Treatment C: Maribavir 400 mg; Test type: Equivalence — A linear mixed-effects model was applied to ln-transformed AUC0-infinity with treatment, period, and sequence as fixed effects, and participant within sequence as a random effect. Point estimates and their associated 90% CIs was constructed for differences between Treatment C versus Treatment A. The point estimates and their associated 90% CIs were then back transformed to provide point estimates and 90% CIs for ratios of Treatment C versus Treatment A; Geometric Mean Ratio (%) = 87.84, 90% CI 2-sided [84.30 to 91.53] — Geometric mean ratio (%) was calculated as 100*(Treatment C / Treatment A)

4. Secondary Outcome: Number of Participants Who Experienced at Least One Treatment-emergent Adverse Event (TEAEs) and Serious TEAEs
Description: TEAEs were defined as adverse events (AEs) with a start date on or after the first dose of the ID, or with a start date before the date of first dose of the ID but increasing in severity after the first dose of the ID. An SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital abnormality or birth defect, an important medical event. Any clinically significant changes from baseline in vital signs, electrocardiograms (ECGs), and clinical laboratory results were reported as TEAEs. Number of participants who experienced at least one TEAEs and serious TEAE were reported.
Time Frame: From start of study drug administration to follow-up (up to Day 18)
Population: The safety set included all participants who received at least 1 dose of maribavir.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Maribavir 400 mg | Treatment B: Maribavir 400 mg | Treatment C: Maribavir 400 mg
Number analyzed (Participants) | 31 | 30 | 31
Participants
  TEAEs | 11 | 10 | 7
  Serious TEAEs | 0 | 0 | 0

5. Secondary Outcome: Number of Participants Based on Severity of TEAEs
Description: Severity of TEAEs were determined by following criteria: Mild: An AE that was usually transient and might require only minimal treatment or therapeutic intervention. The event did not generally interfere with usual activities of daily living; Moderate: An AE that was usually alleviated with additional specific therapeutic intervention. The event interfered with usual activities of daily living, causing discomfort but possessed no significant or permanent risk of harm to the research participant; Severe: An AE that interrupted usual activities of daily living, or significantly affects clinical status, or might require intensive therapeutic intervention. Number of participants based on severity of TEAEs as assessed by the Investigator were reported.
Time Frame: From start of study drug administration to follow-up (up to Day 18)
Population: The safety set included all participants who received at least 1 dose of maribavir.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Maribavir 400 mg | Treatment B: Maribavir 400 mg | Treatment C: Maribavir 400 mg
Number analyzed (Participants) | 31 | 30 | 31
Participants
  Mild | 11 | 10 | 7
  Moderate | 0 | 0 | 0
  Severe | 0 | 0 | 0

6. Secondary Outcome: Number of Participants Based on Causality of TEAEs
Description: The causality relationship of each AE to the ID was assessed using the following categories: Related: An AE that followed a reasonable temporal sequence from administration of a drug (including the course after withdrawal of the drug), or for which a causal relationship was at least a reasonable possibility, that was, the relationship could not be ruled out, although factors other than the drug, such as underlying diseases, complications, concomitant drugs and concurrent treatments, might also be responsible; Not Related: An AE that did not follow a reasonable temporal sequence from administration of a drug and/or that could reasonably be explained by other factors, such as underlying diseases, complications, concomitant medications and concurrent treatments. Number of participants based on causality of TEAEs as assessed by the Investigator were reported.
Time Frame: From start of study drug administration to follow-up (up to Day 18)
Population: The safety set included all participants who received at least 1 dose of maribavir.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Maribavir 400 mg | Treatment B: Maribavir 400 mg | Treatment C: Maribavir 400 mg
Number analyzed (Participants) | 31 | 30 | 31
Participants
  Related TEAEs | 8 | 9 | 7
  Not Related TEAEs | 3 | 1 | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration to follow-up (up to Day 18)
Arm/Group | Treatment A: Maribavir 400 mg | Treatment B: Maribavir 400 mg | Treatment C: Maribavir 400 mg
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 7/31 | 9/30 | 7/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Maribavir 400 mg (N=31) | Treatment B: Maribavir 400 mg (N=30) | Treatment C: Maribavir 400 mg (N=31)
Dysgeusia (Nervous system disorders) | 6 | 8 | 5
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT05382104/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT05382104/SAP_001.pdf